CLINICAL TRIAL: NCT05852873
Title: PAxlovid loNg cOvid-19 pRevention triAl With recruitMent In the Community in Norway
Acronym: PanoramicNOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Oslo University Hospital (Other); University of Oslo (Other); St. Olavs Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC-SE-578741
Record Dates: First submitted 2023-05-08; First posted 2023-05-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Post COVID-19 Condition, Unspecified; SARS-CoV2 Infection; COVID-19
Keywords: Nirmatrelvir ritonavir; Prevention
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Double-blinded placebo-controlleded randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nirmatrelvir-ritonavir (Active Comparator): Participants will receive a standard 5-day treatment course nirmatrelvir plus ritonavir in addition to standard of care. The participants will receive 2 tablets nirmatrelvir 150 mg twice daily and 1 tablet ritonavir 100mg twice daily, both for a duration of 5 days. The tablets have been encapsulated to maintain blinding.
  Interventions: Drug: Nirmatrelvir/ritonavir
- Placebo (Placebo Comparator): Participants in the control arm will receive a 5-day course of placebo tablets in addition to standard of care. The participants will receive 3 tablets twice daily for 5 days. The placebo tablets have the same shape and appearance as the active comparator product. The tablets containing placebo and active comparato have both been encapsulated in the same way to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — Participants in the intervention arm will receive a standard 5-day treatment course Paxlovid (nirmatrelvir plus ritonavir) in addition to standard of care.
  Other Names: Paxlovid tablets
  Arms: Nirmatrelvir-ritonavir
Drug: Placebo — Participants in the control arm will receive a 5-day course of placebo tablets, with the same appearance and quantity, in addition to standard of care.
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare treatment with oral Paxlovid (nirmatrelvir/ritonavir) and placebo for acute COVID-19 as an intervention to prevent long-COVID (post-COVID-19 condition) in adults aged 18-64 years old.

The main question it aims to answer is:

Does treatment with Paxlovid for acute COVID-19 reduce the prevalence of long-COVID compared to placebo.

Participants with acute COVID-19, documented with positive lateral flow test or PCR, within the last 5 days will be randomised to take either Paxlovid or placebo. All participants will receive standard of care in addition. Participants will respond to electronic questionnaires at 14 time points during follow-up. The primary outcome is presence of long-COVID symptoms at 3 months follow-up.

Researchers will compare participants who received Paxlovid and placebo to see if Paxlovid treatment can prevent the occurrence of long-COVID.

DETAILED DESCRIPTION:
PAxlovid loNg cOvid-19 pRevention triAl with recruitMent In the Community in Norway

Background: Despite high uptake of vaccination against COVID-19, the disease remains prevalent in Norway and in many countries around the world, with many patients continuing to experience considerable morbidity and requiring hospital treatment. There is therefore an urgent need to identify treatments for COVID-19 for use in the community early on in the illness that speeds recovery and prevents the need for hospital admission. A considerable burden of long term complications has been reported after COVID (named long COVID) even after home isolation of mild cases, but are particularly associated with more severe disease, and an early therapeutic intervention could potentially also prevent this COVID-19 related morbidity.

Aims and objectives: The study hypothesis is that antiviral treatment for acute Covid can prevent occurrence of persisting symptoms at 3 months and beyond. The primary objective is to assess whether a 5-day course of nirmatrelvir/ritonavir (Paxlovid ®) treatment for patients with acute Covid verified by positive SARS-CoV-2 PCR test result or positive lateral flow test, can reduce the prevalence of persistent symptoms at 3 months compared to placebo. The overall aim of the research is to identify a tool to prevent long COVID, and reduce its burden on society.

Interventions: This is a randomized clinical trial assessing whether healthy adults (P) treated with Paxlovid (I) for acute Covid versus those treated with placebo (C) will have reduced probability of suffering persistent symptoms at 3 months and beyond (O). Participants will be randomized 1:1 to two arms of the trial. Participants in the intervention arm will receive a standard 5-day treatment course Paxlovid (nirmatrelvir plus ritonavir) in addition to standard of care. Participants in the control arm will receive a 5-day course of placebo tablets, with the same appearance and quantity, in addition to standard of care. Participants will be randomised to receive either the antiviral agent Paxlovid (nirmatrelvir plus ritonavir) in addition to standard of care or Placebo plus standard of care.

Eligibility: Participants who meet the following inclusion criteria may be eligible to take part in the trial:

* Symptoms attributable to COVID-19 starting within the past 5 days and ongoing
* A positive PCR SARS-CoV-2 test or a positive lateral flow test. Any positive PCR test or a lateral flow test taken between two days before symptom onset and randomisation qualifies
* Age ≥ 18 years and <65 years
* Participant is able and willing to provide informed consent, and able to comply with all study visits
* Patient not currently admitted to hospital
* No comorbidity which constitutes an indication for active antiviral treatment with Paxlovid as judged by the investigator
* No chronic renal impairment
* No chronic liver disease or liver impairment
* No previous randomisation in the PANORAMIC Norway trial
* Not currently participating in a clinical trial of a therapeutic agent
* Not currently taking Paxlovid
* No known allergy to Paxlovid
* No use of concomitant medication contraindicated for the treatment of Paxlovid
* Not currently pregnant or lactating
* Willingness to take a pregnancy test prior to starting study treatment (Participants of childbearing potential)
* Willingness to use highly effective contraceptive until 7 days after completing Paxlovid (Participants of childbearing potential or have a partner of childbearing potential)

Outcomes: The primary endpoint will be presence of pre-defined symptoms of long COVID at 3 months from randomisation). The secondary outcome will be all-cause, non-elective hospitalisation or death within 28 days of randomisation. Secondary outcomes will further include time to self-reported recovery; participant reported illness severity; duration of symptoms and symptom recurrence; healthcare service use; participant reported household infection rate; safety outcomes and cost-effectiveness outcomes; symptoms and well-being at six months (with determination of proportion with Long Covid) from randomisation. See Table 1 for details of objectives and outcome measures.

Study design: This is a two-arm 1:1 randomized double-blinded placebo-controlled clinical trial. The study is designed to assess whether healthy adults (P) treated with Paxlovid (I) for acute Covid versus those treated with placebo (C) will have reduced probability of suffering persistent symptoms at 3 months and beyond (O). An external statistician will produce a randomization list prior to the start of the trial. At the time of inclusion in the study, study personnel will blindly allocate participants to receive active ingredient or placebo according to the randomization list. All enrolment (screening, eligibility review, informed consent and baseline data) will be conducted by the trial team, with follow-up procedures (electronic diary) conducted remotely with participants or their chosen support person (Study Partner) using the trial website or a telephone call with the trial team. Any hospitalisations and deaths will be recorded.

Recruitment: A central trial team will recruit and allocate participants to the next medication/Placebo number. A participant pack containing Paxlovid or Placebo will be given to the participant or their Study Partner, which is a person appointed by the participant to act on their behalf, for instance to collect study medication at the central study site. During the study period, further recruitment sites and PraksisNett collaboration will be considered.

Data to be recorded: Demographic features including age, gender, comorbidity, allergies, medication history and present medication, COVID vaccine history and previous COVID-19 will be captured at baseline. In the online diary (completed each day for 7 days, weekly for 28 days, and at 3 and 6 months) and during telephone calls, participants or their Study Partners will rate the severity of symptoms including how well they are feeling, record contacts with the health services (including hospital admission), record study medication use, resource use, sick leave, and new infections in the household. Follow-up beyond 28 days after randomisation will be by accessing medical registries and by participant questionnaire for information relevant to the longer-term consequences of COVID-19 at three and six months from randomisation. To investigate the impact of trial interventions on the longer-term effects of COVID-19, we will also remotely follow-up participants, for up to 1 year.

Exploratory subprojects: 1. A subgroup of up to 500 patients will be asked to attend a face-to-face visit or to donate a microbiological or blood sample for the purpose of the study, at 3, 6 and 12 months after inclusion. 2. A smaller group of 100 patients, with and without symptoms at 3 months will be included in a study on brain damage, including neurocognitive, EEG and MRI investigations.

Numbers to be randomised: An estimated maximum of approximately 1000 participants per arm will be required to provide approximately 90% power for detecting a 20% relative reduction in long COVID symptoms in an experimental arm relative to Placebo, based on the assumption of an underlying 30% prevalence of long COVID at 3 months in the placebo arm, and an intervention lowering the long COVID rate to 22%.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms attributable to COVID-19 started within the past 5 days and ongoing
* Positive PCR or lateral flow SARS-CoV-2 test. Any positive PCR test or a lateral flow test taken between two days before symptom onset and randomisation qualifies.
* Age between 18 and 65 years
* Participant is able and willing to provide informed consent
* Willingness to take a pregnancy test prior to starting study treatment (Participants of childbearing potential)

Exclusion Criteria:

* Patients that are not able to comply with all study visits
* Patient currently inpatient at hospital
* Comorbidity which requires active antiviral treatment as judged by the investigator
* Any chronic renal impairment
* Any chronic liver disease or liver impairment
* Previous randomisation in the PANORAMIC Norway trial
* Currently participating in a clinical trial of a therapeutic agent
* Currently taking Paxlovid
* Known allergy to Paxlovid
* Use of concomitant medication contraindicated for the treatment of Paxlovid*
* Pregnant and lactating women
* Participants of childbearing potential (participants who are anatomically and physiologically capable of becoming pregnant), or have a partner of childbearing potential, not willing to use highly effective contraceptive until 7 days after completing Paxlovid.

  * Concomitant medications that are contraindicated for the treatment of Paxlovid
* Medicinal products that are highly dependent on CYP3A for clearance and for which elevated concentrations are associated with serious and/or life-threatening reactions.
* Medicinal products that are potent CYP3A inducers where significantly reduced nirmatrelvir/ritonavir plasma concentrations may be associated with the potential for loss of virologic response and possible resistance. Paxlovid cannot be started immediately after discontinuation of such medicinal products due to the delayed offset of the recently discontinued CYP3A inducer.

More information is available in the study protocol on medicinal products that are contraindicated with concomitant use of Paxlovid.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Symptoms of long-COVID | Change in symptoms from baseline to 3, 6 and 12 months follow-up
  a dichotomous variable for presence of any of the three most important long-COVID symptoms: (i) fatigue, (ii) dyspnea and (iii) cognitive symptoms (defined as memory and/or concentration problems).

SECONDARY OUTCOMES:
Symptoms individually and grouped by organ system | Change in symptoms from baseline to 3, 6, 12 and 24 months follow-up
  All individual symptoms separately, and grouped by systems (systemic symptoms, chest-symptoms, cognitive, other neuropsychiatric symptoms).
Graded responses for symptoms and symptom constellations | Change in symptoms from baseline to 3, 6, 12 and 24 months follow-up
  Graded responses for separate symptoms and symptom constellations, including an ordinal variable graded 0-3 for the presence of the 3 symptoms in the primary outcome.
Risk factors for long-COVID | Up to 24 months
  Analysis of patient characteristics and other factors that may affect the occurrence of long-COVID
Severity of acute disease | 28 days
  Severity of acute disease using an 8-step scale (1 - no limitation of activities, 2 - limitations of activities, not hospitalised, 3 - hospitalised not requiring specific treatment, 4 - hospitalised, requiring medical treatment, but not supplemental oxygen, 5 - need of supplemental oxygen, 6 - need of non-invasive ventilatory support (CPAP, BiPAP), 7 - need ov invasive ventilation, 8 - death
Hospitalisation | 28 days
  Hospitalisation - binary outcome
Severe adverse events | Up to 24 months
  Severe adverse events
Absence from work | Up to 24 months
  Absence from work, full or partial sick leave
Societal costs | Up to 24 months
  Societal cost / economic analysis, including estimated cost of absence from work/school, hospitalizations, deaths, QALYs lost according to EQ-5D-5L, and more
Symptoms of long-COVID | Change in symptoms from baseline to 3, 6 and 12 months follow-up
  a dichotomous variable for presence of any of the three most important long-COVID symptoms: (i) fatigue, (ii) dyspnea and (iii) cognitive symptoms (defined as memory and/or concentration problems).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Langeland, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared with other researchers upon reasonable request, provided patient confidentiality is fully maintained
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion and after the publication of the main outcomes of the trial.
Access Criteria: Individual participant data may be shared with other researchers upon reasonable request, provided patient confidentiality is fully maintained

REFERENCES:
- [Background] McNicoll N, Gagnon J, Rondeau JJ, Ong H, De Lean A. Localization by photoaffinity labeling of natriuretic peptide receptor-A binding domain. Biochemistry. 1996 Oct 1;35(39):12950-6. doi: 10.1021/bi960818q. PMID 8841141
- [Background] Yasin SA, Costa A, Besser GM, Hucks D, Grossman A, Forsling ML. Melatonin and its analogs inhibit the basal and stimulated release of hypothalamic vasopressin and oxytocin in vitro. Endocrinology. 1993 Mar;132(3):1329-36. doi: 10.1210/endo.132.3.8440190.
- [Background] Franke DR, Nuttall KL. Orotic acid in clinical urine specimens by capillary zone electrophoresis using polyvinyl alcohol coated capillaries. J Capillary Electrophor. 1996 Nov-Dec;3(6):309-12. PMID 9384725
- [Background] Boyce ST, Greenhalgh DG, Kagan RJ, Housinger T, Sorrell JM, Childress CP, Rieman M, Warden GD. Skin anatomy and antigen expression after burn wound closure with composite grafts of cultured skin cells and biopolymers. Plast Reconstr Surg. 1993 Apr;91(4):632-41. doi: 10.1097/00006534-199304000-00010. PMID 8446717
- [Background] Stokel-Walker C. The search for antivirals for covid-19. BMJ. 2021 Sep 20;374:n2165. doi: 10.1136/bmj.n2165. No abstract available. PMID 34544682
- [Background] Kim PS, Read SW, Fauci AS. Therapy for Early COVID-19: A Critical Need. JAMA. 2020 Dec 1;324(21):2149-2150. doi: 10.1001/jama.2020.22813. No abstract available. PMID 33175121
- [Background] Dorey G, Dubois L, Prodo de Carvalho LP, Potier P, Dodd RH. Synthetic routes to 4-amino-3-carboxy-beta-carboline derivatives: incidental formation of novel furo[3,4-c]-beta-carbolin-2-ones displaying high affinities for the benzodiazepine receptor. J Med Chem. 1995 Jan 6;38(1):189-98. doi: 10.1021/jm00001a024. PMID 7837230
- [Background] Ghittori S, Maestri L, Maraccini P, Imbriani M. Acetone in urine as biological index of occupational exposure to isopropyl alcohol. Ind Health. 1996;34(4):409-14. doi: 10.2486/indhealth.34.409. PMID 8908851
- [Background] Crandall CS. Prejudice against fat people: ideology and self-interest. J Pers Soc Psychol. 1994 May;66(5):882-94. doi: 10.1037//0022-3514.66.5.882. PMID 8014833
- [Background] Nook TH. In vivo measurement of the keratolytic effect of salicylic acid in three ointment formulations. Br J Dermatol. 1987 Aug;117(2):243-5. doi: 10.1111/j.1365-2133.1987.tb04123.x. PMID 3651343
- [Background] Ertesvag NU, Iversen A, Blomberg B, Ozgumus T, Rijal P, Fjelltveit EB, Cox RJ, Langeland N; Bergen COVID-19 research group. Post COVID-19 condition after delta infection and omicron reinfection in children and adolescents. EBioMedicine. 2023 Jun;92:104599. doi: 10.1016/j.ebiom.2023.104599. Epub 2023 May 5. PMID 37149931
- [Derived] Blomberg B, Myklebust NN, Oppegaard O, Tondel C, Cox RJ, Iversen A, Lehmann ME, Sandvig A, Dahl TB, Valderhaug VD, Szodoray P, Wilhelmsen M, Kirsebom BE, Glambek M, Kaarboe O, Aukrust P, Lie RT, Langeland N. Randomized trial of nirmatrelvir/ritonavir versus placebo for adults with acute COVID-19 to prevent long COVID: PanoramicNOR Trial. Trials. 2025 Nov 6;26(1):477. doi: 10.1186/s13063-025-09226-6. PMID 41199272

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT05852873/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT05852873/SAP_002.pdf